CLINICAL TRIAL: NCT05666609
Title: Fistula-in-ano in Infants and Children: Prospective, Randomized Clinical Trail on the Duration of Non-cutting Seton Placement
Brief Title: Fistula-in-ano in Infants and Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Dr. med. Sonja Diez, Medical Doctor, Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIA2023-7
Record Dates: First submitted 2022-12-18; First posted 2022-12-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Fistula in Ano
MeSH Terms: conditions — Rectal Fistula | interventions — Silicones

STUDY DESIGN:
Intervention Model Description: Group A: duration of placed seton 4 weeks Group B: duration of placed seton 12 weeks
Masking Description: Masking is not possible due to study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 4weeks (Active Comparator): Duration of placed seton 4 weeks
  Interventions: Procedure: placement of non-cutting seton (silicone)
- Group 12weeks (Active Comparator): Duration of placed seton 12 weeks
  Interventions: Procedure: placement of non-cutting seton (silicone)

INTERVENTIONS:
Procedure: placement of non-cutting seton (silicone) — Treatment of Fistula in ano is conducted according to the institution's treatment guidelines. Silicon seton placement is conducted under general anesthesia. Identification of the FIA is secured by the insertion of a bulb-headed lacrimal probe, on which a silicon vessel loop is attached and pulled through the entire fistulous tract. In case of a perianal abscess, drainage and sphincter-sparing debridement is performed followed by secondary wound healing. The loop is ligated loosely outside the anus without any additional tension to the skin. Duration of placed seton is depending on group assignment and is set to either 4 or 12 weeks.

SUMMARY:
In this prospective, randomized trail, duration of non-cutting seton placement in patients with fistula-in-ano is evaluated.

DETAILED DESCRIPTION:
In this prospective, randomized trail, patients are treated in case of fistula-in-ano with non-cutting seton placement. They are then randomized 1:1 in either Group A (duration of placed seton for 4 weeks) or Group B (duration of placed seton for 12 weeks). Patients are participating after informed consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

* any patient with FIA and treatment with non-cutting seton placement in our institution
* regardless of underlying diagnoses
* age 0-18 years

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent fistula in ano | 6 months after initial surgery
Recurrent perianal abscess | 6 months after initial surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Diez, MD, Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Friedrich-Alexander-Universität Erlangen-Nürnberg, Pediatric Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No